CLINICAL TRIAL: NCT05709743
Title: Task Switching Between Positive and Negative Target Templates During Visual Search in Healthy Adults
Brief Title: Task Switching Between Target Templates During Visual Search in Healthy Adults
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Lehigh University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 4R15EY030247-01A1 (NIH)
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Healthy
Keywords: attention; visual search

STUDY DESIGN:
Intervention Model Description: All participants receive each level of visual information (target or distractor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Within-Subjects Attentional Information (Experimental): Within-Subjects, all participants receive all interventions
  Interventions: Behavioral: Experimental: Within-Subjects Attentional Information

INTERVENTIONS:
Behavioral: Experimental: Within-Subjects Attentional Information — Behavioral: Visual Search Information Type (target or distractor information) Participants will have information about targets, distractors, or neither in different trials of the intervention.
  Other Names: Within-Subjects, all participants receive all interventions

SUMMARY:
In this line of research, the researchers having participants engage in task switching between tasks which require a positive (target) template, negative (distractor) template, or neutral (non-informative) template to the cognitive control factors associated with each template type during visual search. This is a basic science study.

DETAILED DESCRIPTION:
The researchers will have participants engage in task switching between tasks which require a positive (target) template, negative (distractor) template, or neutral (non-informative) template to the cognitive control factors associated with each template type during visual search. Looking for impacts of task switching helps to identify the components of the cognitive control system that overlap between different types of attentional templates. This is a basic science study.

ELIGIBILITY:
Inclusion Criteria:

* normal or corrected to normal visual acuity, normal color vision

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2025-02-17 (Estimated); Study Completion 2025-06-17 (Estimated)

PRIMARY OUTCOMES:
Button Press Reaction Time | One day (during testing)
  Speed to respond correctly to the target- after participant finds the target shape on a computer screen, they press a button to indicate what shape they see
Button Press Accuracy | One day (during testing)
  Accuracy of responses to target item (% correct)- the researchers will measure whether the participants presses the correct button which corresponds to the target shape presented on the computer screen or the incorrect button
Eye Movements to Objects on Computer Screen | One day (during testing)
  Proportion (% of total) of eye movements directed to potential targets or distractors, measured with an Eye Link II eye tracker

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Carlisle, PhD, Principal Investigator — Lehigh University
Locations (1):
- Lehigh University, Bethlehem, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The researchers plan to share anonymized subject data on Open Science Framework.
Supporting Information: Study Protocol, SAP
Time Frame: Upon publication.
Access Criteria: Open Science Framework internet access.